CLINICAL TRIAL: NCT06030050
Title: Animal Assisted Intervention for Hemodialysis Outpatients: A Mixed-method Randomized Controlled Trial for Treatment Adherence and Psychosocial Well-being
Brief Title: Animal Assisted Intervention for Hemodialysis Outpatients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was not feasible to conduct.
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: U.S. Renal Care, Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20230396HU
Record Dates: First submitted 2023-08-31; First posted 2023-09-08 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: End-Stage Kidney Disease; Chronic Kidney Failure; Chronic Pain
Keywords: treatment adherence
MeSH Terms: conditions — Kidney Failure, Chronic; Chronic Pain; Treatment Adherence and Compliance

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): Intervention: Animal-assisted intervention (therapy dog visit) Frequency: 2 dog visits per week Duration: each visit is approx 10 mins long, study lasts 20 weeks
  Interventions: Behavioral: Animal-assisted intervention
- Control group (No Intervention): Intervention: NONE - sit in waiting room like usual Frequency: 0 dog visits per week Duration: study lasts 20 weeks

INTERVENTIONS:
Behavioral: Animal-assisted intervention — The AAI is designed to promote patient comfort, uplift mood, and provide an opportunity for socialization. The nature of the dog interaction involves several different components, including but not limited to: petting the dog, talking to the dog, watching the dog do tricks, conversing with the dog handler, and being prompted to discuss any fond memories/stories of their own personal experiences with human-animal interactions. Therapy dogs are trained and certified animals who are leashed at all times and under direct care of their dog handler, NOT companion animals, personal pets, nor emotional support animals.
  Arms: Treatment group

SUMMARY:
The goal of this clinical trial is to understand if and how an animal-assisted intervention [AAI] using therapy dogs can support hemodialysis [HD] patients' treatment adherence and enhance their well-being. The main objectives are:

* Objective 1: Determine if the AAI impacts patients' HD treatment adherence (primary outcome is number of unplanned missed treatments no due to hospitalization).
* Objective 2: Evaluate if the AAI impacts patients' psychosocial well-being (secondary outcomes are stress, pain, mood, QOL).
* Objective 3: Examine potential mechanistic biomarkers that underpin human-animal bonding (hormones tied to stress and bonding). (exploratory aim)
* Objective 4: Understand patients' subjective experiences of the AAI.

Participants will be asked to engage in several research tasks, including:

* assessments
* therapy dog visits
* monthly blood draws
* focus group

Researchers will compare how the treatment group (those who receive 2 dogs visits per week) and the control group (those who receive 0 dog visits per week) to see if the AAI impacts treatment adherence and psychosocial well-being.

DETAILED DESCRIPTION:
This study will take place in one outpatient dialysis clinic. The clinical trial will compare a standardized therapy dog interaction delivered twice weekly (based on pilot study outcomes detailed below) to usual care (e.g., no dog exposure) using a 1:1 randomized, 2-arm design. Subjective patient-reported outcomes [PRO] and routinely-tracked clinic data (e.g., missed visits) will be used. A total of 30 patients will be recruited then randomized 1:1 into 2 arms: control group with 0 dog visits (n = 15) and intervention group with 2 dog visits per week for 20 weeks (n = 15). The AAI is designed to promote patient comfort, uplift mood, and provide an opportunity for socialization. The nature of the dog interaction involves several different components, including but not limited to: petting the dog, talking to the dog, watching the dog do tricks, conversing with the dog handler, and being prompted to discuss any fond memories/stories of their own personal experiences with human-animal interactions. Regarding duration, the dog visits average 10 minutes but will be allowed to vary, and length of dog visits will be tracked. Each team (dog handler + dog) will have an assigned unique ID so that variation in dog is controlled for. This study will utilize trained certified dog handlers to deliver the intervention from reputable local and national pet therapy organizations. All dogs have gone through extensive training and behavioral assessment, will provide proper documentation, liability insurance, and vaccinations. All study procedures take place in the clinic waiting room. Patient-reported outcomes (PRO)s will be collected as pre-post data (before and after dog visit or lobby-as-usual control condition). All PROs will be collected electronically on iPads using REDcap. Regarding treatment adherence data, the clinic routinely tracks missed appointments and will report these metrics directly to research team. Patients will complete assessments 2 times per week for a total of 20 weeks. A short demographic questionnaire will be administered once at the first study visit. Also, patients will also undergo a monthly blood-draw providing 3mL of blood 1 time a month at the same time as their standard of care blood draw. This will be bio-banked in a repository for later ELISA analyses, which will focus on hormones related to stress and bonding (e.g., oxytocin, cortisol); this may provide insight into mechanistic biomarkers underpinning the human-animal bonding process. Lastly, qualitative focus groups with intervention group participants will be conducted post-trial to learn about their subjective experiences of the AAI.

ELIGIBILITY:
Inclusion Criteria:

* current HD patient
* aged 18+,
* English speaking, -≥2 missed HD treatments in the last 90 days.

Exclusion Criteria:

* not an HD patient currently
* aged younger than 18 years old
* lacks proficiency in English speaking and reading
* has only 1 or less missed HD treatments in the last 90 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2024-01 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Treatment adherence | 20 weeks
  Number of unplanned missed hemodialysis treatment sessions not due to hospitalizations

SECONDARY OUTCOMES:
Affective distress | 20 weeks
  Anxiety & depression (PHQ-4). This is 4 items. Total score is determined by adding together the scores of each of the 4 items. Scores are rated as normal (0-2), mild (3-5), moderate (6-8), and severe (9-12). Total score ≥3 for first 2 questions suggests anxiety. Total score ≥3 for last 2 questions suggests depression.
Pain unpleasantness | 20 weeks
  Pain unpleasantness (Numeric Rating Scale 0-10) This is 1 item. higher score means worse pain.
Pain intensity | 20 weeks
  Pain intensity (PROMIS-SF). This is 3 items, score range 3 - 15 (raw scores) , higher scores indicate worse pain.
Stress | 20 weeks
  Subjective psychological stress (Stress symptom scale). 1 item, 5-point likert scale, higher score indicates greater stress.
Dog bonding | 20 weeks
  Human Animal Bond Scale. Emotionality sub-scale (7 items). 5-pt likert scale. Higher scores indicate higher levels of bonding between human and animal.
Companionship | 20 weeks
  Social togetherness (PROMIS-SF companionship). 4 items. 5-pt likert scale. Higher scores indicate higher levels of companionship.
Social Support | 20 weeks
  Emotional support (PROMIS-SF Emotional support). 4 items. 5-pt likert scale. Higher scores indicate higher levels of support.
Perceived subjective Quality of life | 20 weeks
  Perceived overall quality (Kemp QOL scale). 1 item. 7-pt likert scale, higher score indicates better perceived quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Meredith L Stensland, PhD, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (1):
- US Renal Care Dialysis Clinic, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared upon request when study data is analyzed and published in a peer review journal.

REFERENCES:
- See also: Study collaborate website (U.S. Renal Care, Inc.) — https://www.usrenalcare.com/